CLINICAL TRIAL: NCT01868802
Title: Ketamine for Treatment-resistant Depression: A Multicentric Clinical Trial in Mexican Population
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul J. Lamothe (Other)
Responsible Party: Sponsor-Investigator, Paul J. Lamothe, Chief of the Research Department, Neurological Center., American British Cowdray Medical Center
Organization: American British Cowdray Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABC KET-DRT-01-2013
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Depressive Disorder,; Treatment-Resistant Depression
Keywords: Ketamine; Depression; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine treated (Experimental)
  Interventions: Drug: Ketamine
- Control, placebo treated (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — A single dose of 0.5mg/kg intravenous ketamine infusion will be administered over 40 minutes.
  Other Names: Ketalar
  Arms: Ketamine treated
Drug: Placebo — Saline at 0.9% intravenous infusion will be administered over 40 minutes.
  Arms: Control, placebo treated

SUMMARY:
A randomized multicentric parallel arms study involving the use of ketamine for treatment-resistant depression will be held at three national health provider clinics in the Mexican population. The purpose of this study is to determine whether clinical response seen in previous studies is replicable in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old
* Mayor Depressive Disorder Diagnosis based on DSM-IV TR.
* Classification of MDD as treatment-resistant.
* No brain structural abnormalities as evidenced by an MRI scan.
* Signed acceptance of Informed Consent.

Exclusion Criteria:

* Other psychiatric diagnosis apart from MDD.
* Substance abuse or dependence (prior or during study).
* Pregnancy.
* Congestive heart disease.
* Personal history of psychosis.
* First-degree relative with history of psychosis.
* Glaucoma.
* Present neurological disease.
* High blood or pulmonary artery pressure.
* Declining the signing of the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline HDRS Score | 20 minutes before and 40 minutes after ketamine infusion.
  The Hamilton Depression Rating Scale (HDRS) baseline score will be measured 20 minutes before ketamine infusion. After 40 minutes post-infusion, a second HDRS score will be obtained.
Daily change in HDRS post-ketamine infusion. | 1,2,3,4,5,6 and 7. Days after ketamine infusion
  On a daily basis, from day 1-7 post-ketamine infusion, changes in HDRS score will be measured during the daily psychiatric evaluation.

SECONDARY OUTCOMES:
Baseline blood pressure (BP). | 20 minutes before ketamine infusion.
  Baseline BP will be measured during the physical examination 20 minutes before ketamine infusion.
Changes from baseline in blood pressure (BP) | every 5 minutes in a 300 minutes period
  BP will be monitored continuously for a 4-hour period. BP assessments will be taken every five minutes for the period mentioned. The assessment will start 20 minutes before ketamine administration and will finish 4hrs after starting.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Lamothe, M.D., Principal Investigator — American British Cowdray Medical Center; David N Lopez-Garza, M.D., Study Director — American British Cowdray Medical Center; Manuel Ruiz-Alvarez, M.D., Principal Investigator — American British Cowdray Medical Center
Locations (1):
- ABC Neurological Center, Mexico City, Mexico City, Mexico